CLINICAL TRIAL: NCT04856722
Title: Mini-PNL, RIRS, and ESWL for Treatment of Medium-Sized, High-Density, Non-Lower Pole, Renal Stones: A Prospective, Randomized, Comparative Study
Brief Title: Mini-PNL, RIRS, and ESWL for Treatment of Medium-Sized, High-Density, Non-Lower Pole, Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor of Urology and Andrology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uro_Azhar_11_021
Record Dates: First submitted 2021-04-17; First posted 2021-04-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-02

CONDITIONS: Renal Stone; Percutaneous Nephrolithotomy; Retrograde Intrarenal Surgery; Extracorporeal Shockwave Lithotripsy
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mini-PNL group (Experimental): In which PCNL will be performed using miniature nephroscope
  Interventions: Procedure: mini-PNL
- RIRS group (Experimental): In which RIRS will be performed using a flexible ureteroscope
  Interventions: Procedure: RIRS
- SWL group (Experimental): In which extracorporeal shock wave lithotripsy will be performed using Dornier lithotripter SII
  Interventions: Procedure: SWL

INTERVENTIONS:
Procedure: mini-PNL — PCNL using miniature nephroscope. The procedure will be performed under general or regional anaesthesia under fluoroscopy guidance.
  Arms: mini-PNL group
Procedure: RIRS — RIRS using flexible ureteroscope. The procedure will be performed under general or regional anaesthesia under fluoroscopy guidance. Holmium Laser lithotripter will be used for stone fragmentation.
  Arms: RIRS group
Procedure: SWL — SWL using Dornier SII lithotripter. the procedure will be performed under sedoanalgesia, and fluoroscopy will be used for stone localization; for a maximum of 3 SWL session.
  Arms: SWL group

SUMMARY:
The optimal management of medium-sized renal stones remains quite challenging and continues to be contested. In the present study, the investigators will compare mini-PNL, RIRS and SWL in the treatment of non- lower pole, medium size, high dense renal stones regarding the stone-free rate, the safety of the procedures, cost, and patients' and surgeon's satisfaction. Eligible patients will be randomly allocated into three equal groups (mini-PNL, RIRS, and SWL). Postoperative, patients will be followed-up by regularly for 3 months. The study parameters will be compared between groups.

DETAILED DESCRIPTION:
The treatment options for renal stones 10-20 mm include either extracorporeal shock wave lithotripsy (SWL) or endourology (retrograde intrarenal surgery (RIRS) and percutaneous nephrolithotomy (PNL).

SWL is an attractive treatment option for renal stones because it is non-invasive and more acceptable for the patient and can be done under analgesia, sedation, or minimal anaesthesia. However, the limitation of SWL includes a relatively lower stone-free rate (SFR) and the need for repeated sessions and auxiliary procedures. The SFR after SWL is affected by several factors, including body mass index (BMI), stone size, intrarenal stone location, skin-to-stone distance (SSD), and stone density.

The EAU guidelines put endourology and SWL as two equal options in medium-sized non-lower pole renal stones and did not give special attention to the stone density, which is an important predictor for SWL outcome. Several studies reported that the number of SWL sessions increased with increased stone attenuation value (SAV) and SFR decreased significantly in high-density renal stone.

PNL and RIRS have good SFR compared to SWL but might entail a significant risk of morbidity. The improved fURS instrumentation and lithotripsy technology, and development of the miniaturized PNL technique, may lower the procedure-related complications and mPNL and RIRS an alternative and excellent option for medium-sized and even large renal stones The investigators hypothesize that addressing the stone density factor may give a clear recommendation for medium-sized, high-density renal stones. They expected the superiority for either mPNL or RIRS, regarding SFR, without increased morbidity.

The study aims to compare the outcome of mPNL, RIRS, and SWL for treatment of non-lower pole, high-density renal stones of 10 to 20 mm size.

The study will include adult patients with non-lower pole, high-density (>1000 HU) renal stones of 10 to 20 mm size.

Pre-operatively, patients will be evaluated by medical history taking, physical examination. urinalysis, urine culture, complete blood cell count (CBC), liver function tests, coagulation profile, blood urea nitrogen (BUN), serum creatinine, plain abdominal X-ray and computed tomography for urinary tract (CT-UT), Eligible patients will be randomly divided into 3 equal groups. PNL group, in which PNL procedures will be performed using miniature nephroscope, RIRS group, in which RIRS will be performed using flexible ureteroscope and SWL group, in which SWL procedures will be performed using Dornier Lithotripter.

post-operatively, patients will be followed up regularly, for 3 months. The SFR, complication rate, cost, patients' and surgeon's satisfaction will be evaluated and compared between the three groups using the appropriate statistical tests and analytical program.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (both genders)
* Single non-lower pole renal stone.
* Stone size: 10-20 mm.
* Stone density: > 1000 HU.

Exclusion Criteria:

* Pregnant women.
* Morbid obesity.
* Severe orthopaedic deformities.
* Co-morbidities precluding general anaesthesia or prone positioning.
* Uncorrectable coagulation disorders.
* Active urinary tract infection (UTI).
* Stone in a calyceal diverticulum.
* Abnormal renal anatomy.
* Urinary tract obstruction distal to the stone.
* Concomitant pathology that needs intervention in the same setting.
* Advanced hydronephrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Stone-free rate | as detected by non-contrasted computed tomography 3 months after the intervention procedures.
  Stone free status is defined as no residual renal stone or residual fragment(s) less than 4 mm size.
Complication rate | up to 3 months.
  intra- and post-operative complications

SECONDARY OUTCOMES:
Cost of treatment | throughout the study procedure, up to 3 months post-operative.
  The cost of each treatment methods will be estimated, Including the devices, disposable instruments, operating room, bed stay, imaging, laboratory, medications, retreatment and ancillary procedures.
Patients satisfaction | throughout the study procedure, up to 3 months post-operative
  A 5-point scale will be used to assess satisfaction, where 1 is unsatisfied and 5 fully satisfied.
Surgeon's satisfaction. | throughout the study procedure, up to 3 months post-operative
  A 5-point scale will be used to assess satisfaction, where 1 is unsatisfied and 5 fully satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Abul-fotouh Ahmed, MD, Principal Investigator — Al-Azhar University Hospitals, Cairo, Egypt
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed AF, Raafat M, ElDamanhory H, Abdelazim H, Soliman A, ElShazly A, Hindawy M, Anwar M, Algammal M, Soliman A, Daoud A. Prospective randomized trial comparing mini-percutaneous nephrolithotomy, retrograde intrarenal surgery, and shock wave lithotripsy for treatment of medium-sized high-density renal stones. Int Urol Nephrol. 2025 Dec 12. doi: 10.1007/s11255-025-04928-x. Online ahead of print. PMID 41385038